CLINICAL TRIAL: NCT07048743
Title: Psilocybin-assisted Existential, Attachment and Relational (PEARL) Therapy for Caregivers of Patients With Advanced Cancer: A Phase II Open-Label Trial
Brief Title: Psilocybin-assisted Existential, Attachment and RelationaL (PEARL) Therapy for Caregivers of Patients With Advanced Cancer
Acronym: PEARL-C1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PEARL-C1
Record Dates: First submitted 2025-06-04; First posted 2025-07-02 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Caregiver Distress
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PEARL Therapy (Experimental)
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Single high-dose (25mg) capsule of psilocybin taken orally in the context of Psilocybin-assisted Existential, Attachment and RelationaL (PEARL) therapy

SUMMARY:
The PEARL-C1 trial is a phase II open-label trial. Participants will receive a single high-dose (25 mg) of psilocybin in the context of Psilocybin-assisted Existential, Attachment and RelationaL (PEARL) therapy.

DETAILED DESCRIPTION:
Caregivers of patients with advanced cancer often experience high levels of distress but there is currently little evidence-based guidance on how to help caregivers who experience depression, anxiety, anticipatory grief, spiritual suffering, caregiving burden and/or impaired quality of life. Over the past decade, research has shown that psychotherapies incorporating existential, attachment and relational approaches can address the specific needs and challenges of the advanced cancer population and thus help to reduce related distress. Simultaneously, recent research has shown that psilocybin-assisted psychotherapy, in which an individual ingests the psychoactive drug within a carefully monitored therapy, can reduce end-of-life distress and greatly benefit those with advanced disease. The multidisciplinary team has combined these two evidence-based approaches into Psilocybin-assisted Existential, Attachment and RelationaL (PEARL) therapy. PEARL therapy combines elements from psilocybin-assisted psychotherapy, including preparatory therapy sessions, a high-dose drug session, and integration sessions, with important elements from manualized individual psychotherapies designed for patients and their families facing advanced cancer. This study will assess the feasibility, acceptability, and safety of PEARL therapy among caregivers of patients with advanced cancer. This study will contribute to the growing research around the efficacy of psychedelic-assisted therapies for the psychological distress associated with advanced disease and mortality. This type of therapy has the potential to improve quality of life among caregivers of those with advanced disease, to build upon previous findings to help outline the necessary components of therapy, and to inform public policy and clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Participant must reside in Ontario, Canada.
* Ability to speak and read English (participant to provide written informed consent and participate in PEARL intervention, as determined by study personnel).
* No cognitive impairment indicated in medical record or by the primary care physician.
* Primary or significant caregiver of a patient with advanced cancer enrolled in a companion trial of PEARL for patients with advanced cancer or caregiver of a patient receiving psilocybin-therapy through the Special Access Program (SAP) at University Health Network (UHN); such patients will have been recruited from psychosocial oncology or palliative care clinics at Princess Margaret (study physicians to assess appropriateness of inclusion and whether treatment will support the family system).
* At least mild anxiety or depression symptoms, defined as a score of >5 on the General Anxiety Disorder-7 (GAD-7) or >8 on the Patient Health Questionnaire-9 (PHQ-9).
* Interest in and ability to participate in and complete the PEARL intervention and protocol as outlined.
* Normal hepatic functioning as determined by prior medical history or/and screening bloodwork (international normalized ratio [INR]<1.5, aspartate aminotransferase [AST]/alanine transaminase [ALT] < 2x upper limit of normal, normal range bilirubin, platelets ≥150).
* Normal renal functioning as determined by prior medical history or/and screening bloodwork (estimated glomerular filtration rate [eGFR]>45).
* Participants who are sexually active and could become pregnant or inseminate a partner must be using one method of highly effective contraception (hormonal contraceptives (e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device (IUD) or intrauterine system (IUS); vasectomy or tubal ligation). Alternatively, they may use a combination of two or more effective methods of contraception which include male condom, female condom, cervical cap, diaphragm, or contraceptive sponge. These acceptable methods of contraception must be used prior to study entry, during study participation, and for the duration of the study.
* For participants of child-bearing potential, a negative serum pregnancy test result is required at screening. A urine pregnancy test will be administered on the morning of psilocybin administration for applicable participants. Participants cannot be pregnant or nursing through the duration of the study.
* If using prescribed medications or other substances, participants must agree to refrain from taking them if instructed by study investigators. These include:

  * not using any non-prescription medication, nutritional supplement, or herbal supplement except when approved by the treatment team (exceptions will be evaluated by the Sponsor-Investigator and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals).
  * not using nicotine for at least 2 hours before psilocybin administration, and not again until approximately 7 hours after psilocybin administration.
  * consuming approximately the same amount of caffeine-containing beverages (e.g., coffee, tea) that they consumes on a usual morning before arriving at the treatment centre for the psilocybin session day.
  * not taking any as needed medications on the mornings of psilocybin sessions (with the exception of daily and as needed opioid pain medication).
  * refraining from using any psychoactive drugs, including alcoholic beverages, within 24 hours of the psilocybin administration.
* Participants must have a responsible individual to drive them after the dosing session to where they are staying (home, hotel or another location) and to accompany/attend to them because psilocybin may affect their alertness and concentration on the evening of the dosing session.
* Participants must agree not to drive or operate machinery for at least 24 hours after dose administration.
* The therapist involved in the participant's psilocybin dosing session and/or the principal investigators will provide their phone number, in advance of the session, to the participant, in case the participant needs to reach them for emergency support in the 24 hours following the psilocybin dosing session. Because the therapists will change from participant to participant, the study team cannot provide the same emergency phone number to every study participant.

Exclusion Criteria:

* A history of past intolerability to psilocybin or other psychedelics.
* Past/present psychiatric diagnoses of bipolar disorder, any psychotic disorder, active substance use disorders, or dementia.

  a. Participants may have current mild alcohol or cannabis use disorder (meets 3 of 11 diagnostic criteria per The Diagnostic and Statistical Manual of Mental Illnesses [DSM-5]) or moderate alcohol or cannabis use disorder in early remission for the 3 months prior to enrollment (meets 5 of 11 diagnostic criteria per DSM-5).
* Clinically significant suicidal ideation either currently or within the past 6 months, as judged by study clinicians.
* Participant under the age of 30 years who has a first degree relative with a primary psychotic disorder.
* Other personal circumstances or behaviour judged to be incompatible with establishment of rapport or safe exposure to psilocybin.
* Severe hypertension (defined as systolic blood pressure >140 or diastolic pressure >90) based on two readings on the same day. If the second reading remains over 140/90 the participant can be brought in for another reading on a different day. Participants can be re-screened for participation once blood pressure is adequately controlled.
* Hepatic dysfunction (history of cirrhosis and/or abnormal parameters [INR>1.5, elevated AST/ALT 2x upper limit, elevated bilirubin, platelets < 150]) or liver failure, defined as clinical diagnosis of liver fibrosis, cirrhosis of the liver, or advanced liver disease.
* Cardiovascular conditions including uncontrolled hypertension, heart failure (defined as class IV of the New York Heart Association classification), angina, a clinically significant electrocardiogram [ECG] abnormality (e.g., atrial fibrillation without rate control, prolonged Corrected QT Interval (QTc) defined as > 450ms for males or > 470ms for females), transient ischemic attack in the last six months, stroke, peripheral or pulmonary vascular disease (no active claudication).
* Uncontrolled epilepsy or history of seizures.
* Diabetes with inability to skip a meal (lunch), requiring administration of medication more than twice daily, or symptomatic hypoglycemia within the prior 30 days.
* GI bleed in last 6 months.
* Use of other investigational agents that would be inappropriate to take with psilocybin in the judgement of the investigator, psychoactive prescription medications (e.g., benzodiazepines, lithium, SSRIs), medications having a pharmacological effect on serotonin-2a (5-HT2A) receptors (e.g., olanzapine, mirtazapine, or trazodone), medications that are monoamine oxidase (MAO) inhibitors, any potent metabolic inducers (e.g. rifamycin, rifampin, rifabutin, rifapentine, carbamazepine, phenytoin, phenobarbital, nevirapine, efavirenz, Taxol, dexamethasone, St John's wort) or inhibitors (e.g. HIV protease inhibitors, itraconazole, ketoconazole, erythromycin, clarithromycin, troleandomycin). Note: Inhibitors of UGT1A9 and 1A10 may increase systemic psilocin exposure (i.e., the Cmax and AUC) of psilocin and should be discontinued at least five half-lives prior to the administration of psilocybin. Similarly, aldehyde or alcohol dehydrogenase inhibitors should be discontinued at least 5 half-lives prior to the dose of psilocybin.

In suitable participants, contraindicated medications may be tapered by a study physician between study enrolment and the psilocybin session when it is deemed safe to do so and in coordination with the prescribing physician. A safe and appropriate tapering regimen will then be developed based on the particular medication, on a case-by-case basis. If taking an MAO inhibitor, the psilocybin session will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose. Participants prescribed opioids will be allowed to take their usual dose regimen for analgesia, including the use of as needed analgesic medications on psilocybin session days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-02 (Estimated); Primary Completion 2027-12-02 (Estimated); Study Completion 2027-12-02 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility as assessed by the number of caregivers who consent/number of caregivers who meet eligibility criteria. | 30 months
  Used to assess feasibility of PEARL therapy.
Retention feasibility as assessed by the number of caregivers completing primary endpoint measures/number of caregivers consented. | 30 months
  Used to assess feasibility of PEARL therapy.
Adherence feasibility as assessed by the number of caregivers completing all PEARL sessions/number of caregivers consented. | 30 months
  Used to assess feasibility of PEARL therapy.
Acceptability of PEARL therapy from the perspective of the caregivers of patients with advanced cancer obtained through qualitative interviews. | 30 months
  Participants will be interviewed regarding their experiences with PEARL, including acceptability and perceived positive and negative effects of the intervention, with a semi-structured interview guide.
Safety of PEARL therapy. | 30 months
  Safety will be assessed throughout the trial. Adverse events (AEs) attributed to psilocybin will be monitored for and recorded after the psilocybin session. This study will use CTCAE v5.0 to assess AEs.
  Serious adverse events (SAEs) will be tracked until study completion and will be defined as any adverse drug experience that: results in death; that is life-threatening (i.e. any AE that places the participant, in the view of the investigators, at immediate risk of death from the reaction as it occurs); requires hospital admission; results in persistent or significant disability (i.e. a substantial disruption of a person's ability to conduct normal life functions); or may jeopardize the participant or necessitate medical intervention to prevent one of the aforementioned criteria.

SECONDARY OUTCOMES:
Caregiver perspectives on the clinical relevance of potential PEARL therapy outcomes: Anxiety symptoms as assessed with the GAD-7. | 30 months
  The Generalized Anxiety Disorder-7 (GAD-7) is a 7-item self-report scale used to screen for and measure anxiety symptoms. Total score range is 0 to 21. Higher scores indicate higher levels of anxiety.
Caregiver perspectives on the clinical relevance of potential PEARL therapy outcomes: Depressive symptoms as assessed with the PHQ-9. | 30 months
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report scale measuring depressive symptoms. Total score range is 0 to 27. Higher scores indicate greater severity of depression.
Caregiver perspectives on the clinical relevance of potential PEARL therapy outcomes: Broad quality of life construct for family members of patients with serious illness as assessed with the QUAL-E (Fam). | 30 months
  The Quality of Life at the End of Life Measure - Family experience (QUAL-E (Fam)) is a 17-item measure that includes subscales assessing symptom impact, relationship with health care provider, completion, and preparation. For symptom impact, score range is 4 to 20, with higher scores reflecting greater symptom control; for the relationship with healthcare provider, score range is 1 to 5, with lower scores reflecting a better relationship with healthcare providers; for completion, score range is 1 to 5, with lower scores reflecting a greater sense of completion in their relationship with the patient; and for preparation, score range is 4 to 20, with lower scores reflecting greater sense of preparation.
Patient perspectives on the clinical relevance of potential PEARL therapy outcomes: Anticipatory grief as assessed with the AGS. | 30 months
  The Anticipatory Grief Scale (AGS) is a 27-item self-report measure of grief before loss in family caregivers. Total score range is 27 to 135. Higher scores indicate higher levels of anticipatory grief.
Caregiver perspectives on the clinical relevance of potential PEARL therapy outcomes: Subjective burden as assessed with the short version of the BSFC-s. | 30 months
  The short version of the Burden Scale for Family Caregivers (BSFC-s) is a 10-item self-report scale designed to measure the subjective burden of family caregivers. Total score range is 0 to 30. Higher scores indicate greater caregiver burden.
Caregiver perspectives on the clinical relevance of potential PEARL therapy outcomes: Overall measure of spiritual well-being, meaning/peace and faith as assessed with the FACIT-Sp. | 30 months
  The Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being (FACIT-Sp) is a 12-item scale designed to measure important aspects of spirituality including sense of meaning in one's life, harmony, peacefulness and a sense of comfort and strength from one's faith. Total score range is 0 to 48. Higher scores indicate higher spiritual well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hales, MD, PhD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braun M, Mikulincer M, Rydall A, Walsh A, Rodin G. Hidden morbidity in cancer: spouse caregivers. J Clin Oncol. 2007 Oct 20;25(30):4829-34. doi: 10.1200/JCO.2006.10.0909. PMID 17947732
- [Background] Burton LC, Newsom JT, Schulz R, Hirsch CH, German PS. Preventive health behaviors among spousal caregivers. Prev Med. 1997 Mar-Apr;26(2):162-9. doi: 10.1006/pmed.1996.0129. PMID 9085384
- [Background] Glajchen M. The emerging role and needs of family caregivers in cancer care. J Support Oncol. 2004 Mar-Apr;2(2):145-55. PMID 15328817
- [Background] Grunfeld E, Coyle D, Whelan T, Clinch J, Reyno L, Earle CC, Willan A, Viola R, Coristine M, Janz T, Glossop R. Family caregiver burden: results of a longitudinal study of breast cancer patients and their principal caregivers. CMAJ. 2004 Jun 8;170(12):1795-801. doi: 10.1503/cmaj.1031205. PMID 15184333
- [Background] Hales S, Chiu A, Husain A, Braun M, Rydall A, Gagliese L, Zimmermann C, Rodin G. The quality of dying and death in cancer and its relationship to palliative care and place of death. J Pain Symptom Manage. 2014 Nov;48(5):839-51. doi: 10.1016/j.jpainsymman.2013.12.240. Epub 2014 Apr 3. PMID 24703943
- [Background] Holm M, Alvariza A, Furst CJ, Ohlen J, Arestedt K. Psychometric evaluation of the anticipatory grief scale in a sample of family caregivers in the context of palliative care. Health Qual Life Outcomes. 2019 Mar 5;17(1):42. doi: 10.1186/s12955-019-1110-4. PMID 30837000
- [Background] Johansson AK, Grimby A. Anticipatory grief among close relatives of patients in hospice and palliative wards. Am J Hosp Palliat Care. 2012 Mar;29(2):134-8. doi: 10.1177/1049909111409021. Epub 2011 May 19. PMID 21596732
- [Background] Kershaw T, Ellis KR, Yoon H, Schafenacker A, Katapodi M, Northouse L. The Interdependence of Advanced Cancer Patients' and Their Family Caregivers' Mental Health, Physical Health, and Self-Efficacy over Time. Ann Behav Med. 2015 Dec;49(6):901-11. doi: 10.1007/s12160-015-9743-y. PMID 26489843
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Nissim RS, Hales S. Caring for the Family Caregiver: Development of a Caregiver Clinic at a Cancer Hospital as Standard of Care. J Clin Psychol Med Settings. 2023 Mar;30(1):111-118. doi: 10.1007/s10880-022-09891-8. Epub 2022 Jun 14. PMID 35699840
- [Background] Nissim, R., Hales, S., Zimmermann, C., Deckert, A., Edwards, B., & Rodin, G. (2017). Supporting Family Caregivers of Advanced Cancer Patients: A Focus Group Study. Family Relations, 66(5), 867-879
- [Background] Pendergrass A, Malnis C, Graf U, Engel S, Graessel E. Screening for caregivers at risk: Extended validation of the short version of the Burden Scale for Family Caregivers (BSFC-s) with a valid classification system for caregivers caring for an older person at home. BMC Health Serv Res. 2018 Apr 2;18(1):229. doi: 10.1186/s12913-018-3047-4. PMID 29609600
- [Background] Peterman AH, Fitchett G, Brady MJ, Hernandez L, Cella D. Measuring spiritual well-being in people with cancer: the functional assessment of chronic illness therapy--Spiritual Well-being Scale (FACIT-Sp). Ann Behav Med. 2002 Winter;24(1):49-58. doi: 10.1207/S15324796ABM2401_06. PMID 12008794
- [Background] Pitceathly C, Maguire P. The psychological impact of cancer on patients' partners and other key relatives: a review. Eur J Cancer. 2003 Jul;39(11):1517-24. doi: 10.1016/s0959-8049(03)00309-5. PMID 12855257
- [Background] Reinhard SC, Given B, Petlick NH, Bemis A. Supporting Family Caregivers in Providing Care. In: Hughes RG, editor. Patient Safety and Quality: An Evidence-Based Handbook for Nurses. Rockville (MD): Agency for Healthcare Research and Quality (US); 2008 Apr. Chapter 14. Available from http://www.ncbi.nlm.nih.gov/books/NBK2665/ PMID 21328765
- [Background] Rosa WE, Sager Z, Miller M, Bernstein I, Doerner Rinaldi A, Addicott K, Ljuslin M, Adrian C, Back AL, Beachy J, Bossis AP, Breitbart WS, Cosimano MP, Fischer SM, Guss J, Knighton E, Phelps J, Richards BD, Richards WA, Tulsky JA, Williams MT, Beaussant Y. Top Ten Tips Palliative Care Clinicians Should Know About Psychedelic-Assisted Therapy in the Context of Serious Illness. J Palliat Med. 2022 Aug;25(8):1273-1281. doi: 10.1089/jpm.2022.0036. Epub 2022 Mar 14. PMID 35285721
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Steinhauser KE, Voils CI, Bosworth HB, Tulsky JA. Validation of a measure of family experience of patients with serious illness: the QUAL-E (Fam). J Pain Symptom Manage. 2014 Dec;48(6):1168-81. doi: 10.1016/j.jpainsymman.2014.04.006. Epub 2014 May 22. PMID 24858740
- [Background] Theut SK, Jordan L, Ross LA, Deutsch SI. Caregiver's anticipatory grief in dementia: a pilot study. Int J Aging Hum Dev. 1991;33(2):113-8. doi: 10.2190/4KYG-J2E1-5KEM-LEBA. PMID 1955206